CLINICAL TRIAL: NCT01456221
Title: The Impact of Using omega3 Long-chain Polyunsaturated Fatty Acids in Weight Loss and Insulin Resistance in Obese Adolescents
Brief Title: Intervention Study With Omega-3 Fatty Acids for Weight Loss and Insulin Resistance in Adolescents
Acronym: O3WLIRADOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mardia Guadalupe Lopez Alarcon, Doctor, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-2011-785-037
Record Dates: First submitted 2011-10-12; First posted 2011-10-20 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin resistance; Omega3 long chain polyunsaturated fatty acids
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Docosahexaenoic Acids; Maxepa; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega 3 and an hypocaloric diet (Experimental): Participants will receive a supplement containing omega 3: Docosahexaenoic acid (DHA) and EPA fatty acids together with an hypocaloric diet.
  Interventions: Dietary Supplement: Omega3 and an hypocaloric diet.
- Placebo (Placebo Comparator): Participants will receive a supplement containing sunflower oil with an hypocaloric diet.
  Interventions: Dietary Supplement: Sunflower oil with an hypocaloric diet.

INTERVENTIONS:
Dietary Supplement: Omega3 and an hypocaloric diet. — Thirty caps with the supplement will be provided every mo during three mo. Supplement will be administered as gel caps containing 1.1 g of DHA and EPA (®MaxEpa, Merck Laboratory) Hypocaloric diet will start at admission and will continue during the six months of follow-up. It will consist in providing a personalized diet including: a) reduction of 700 Kcal from the usual diet considering lipids and carbohydrates, b) increasing fruits and vegetables intake up to six portions daily each, and c) incrementing the intake of fiber to 30 g a day through the inclusion of whole grains.
  Other Names: DHA and EPA fatty acids; Docosahexaenoic fatty acid; Eicosapentaenoic fatty acid; ®MaxEpa, Merck Laboratory
  Arms: omega 3 and an hypocaloric diet
Dietary Supplement: Sunflower oil with an hypocaloric diet. — Thirty caps with the placebo will be provided every mo during three mo. Placebo will be administered as gel caps containing 1g of sunflower oil, which is omega-3 free, and is not expected to produce anti-inflammatory or insulin sensitivity effects. Hypocaloric diet will start at admission and will continue during the six months of follow-up. It will consist in providing a personalized diet including: a) reduction of 700 Kcal from the usual diet considering lipids and carbohydrates, b) increasing fruits and vegetables intake up to six portions daily each, and c) incrementing the intake of fiber to 30 g a day through the inclusion of whole grains.
  Other Names: Sunflower oil
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if a supplement containing omega-3 long chain polyunsaturated fatty acids for three months reduce obesity and insulin resistance to obese adolescents if administered together with a hypocaloric diet.

DETAILED DESCRIPTION:
Background: In 2006, the prevalence of overweight and obesity combined in scholar and adolescents in Mexico was 26% and 31% respectively, which represents more than double of that reported in year 2000. Together with such increments in the obesity rates, it was observed similar increases in the incidence of other metabolic conditions such as insulin resistance (IR). In a very simplistic manner, it seems that the link between obesity and IR is a chronic inflammatory status because the adipose tissue-derived inflammatory molecules interfere with the uptake of fatty acids and glucose in peripheral tissues.

On the other hand, it is accepted that the long-chain polyunsaturated fatty acids (LCPUFA) omega-3 exhibit anti-inflammatory properties. In addition, it has been also demonstrated the beneficial effect exerted by such fatty acids on insulin sensitivity, and in stabilizing the weight lost achieved with hypocaloric diets.

At present, the prevalence of overweight and obesity combined are in the range of 41-43% in the adolescent population that attend the four areas of influence of the Mexican Institute of Social Security (IMSS) in Mexico City. Interventions addressed to improve the nutritional status of these groups of age are expected to impact the risk for IR and its associated co-morbidities.

Objective: To evaluate the impact of supplementation with LCPUFA omega-3, together with a dietary strategy, on obesity and insulin resistance in a sample of obese adolescents attended in the IMSS.

Methods: In a randomized clinical design, 300 obese individuals, 12-18 years old, will be selected. At selection, individuals will be randomly assigned to receive daily a capsule with 1.1 g LCPUFA omega-3 during three mo together with a hypocaloric diet which follows the World Health Organization (WHO) recommendations (D+O3), or to receive daily a capsule with 1.0 g sunflower oil and a similar diet (P+D). After randomization, dietary information (24h-recall and FFQ), anthropometric measurements, and peripheral blood samples, will be obtained. Blood samples will be used to determine fasting plasma glucose and insulin, and erythrocytes fatty acid profile; such determinations will be repeated at three and six mo of follow-up. Anthropometry and 24 h-recalls will be repeated monthly.

For follow-up, studied subjects will be evaluated monthly to deliver capsules and to check for dietary adherence. Treatments will be administered during three months and the follow-up will continue throughout six months. At the end of the follow-up it is expect that the D+O3 group will present: a) higher decreases in mean weight and body mass index (BMI), b) greater decreases in the mean fasting insulin concentration, homeostasis model assessment (HOMA) index, and IR frequency, c) longer duration of weight lost.

Statistical analyses: Student and paired-t test will be used for inter and intra group comparisons respectively. Logistic regression models and repeated measures analyses will be conducted to evaluate the effect of treatments, adjusting by diet and weight loss, as well as by confounders such as puberty and treatment adherence.

Infrastructure: The Unit of Research in Medical Nutrition owes the equipment needed to conduct the laboratory determinations proposed in this research, as well as the personnel qualified to conduct, monitor, analyze and evaluate data from field investigation, specially that related to obesity and IR.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 18 years,
* Male and female
* Body mass Index (BMI) above the 95 percentile of the National Center for Health Statistics (NCHS) reference
* Informed consent form signed by both parents or legal guardian.

Exclusion Criteria:

* Those diagnosed as with Diabetes Mellitus Type 2 (DMT2), Cardiovascular disease (CVD) or kidney disease
* Those who are allergic to fish.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 366 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardia Lopez-Alarcon, PhD, Principal Investigator — Unit for Medical Research in Nutrition, Pediatric Hospital CMN "Siglo XXI"
Locations (1):
- Unit or research in Medical Nutrition, Pediatric Hospital CMN "Siglo XXI", Instituto Mexicano del Seguro Social, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents were recruited between July 2012 and December 2015, from three Family Medicine clinics of the Mexican Institute of Social Security (IMSS) in Mexico City.
Period: Overall Study
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
Started | 183 | 183
Completed | 119 | 126
Not Completed | 64 | 57
Not completed — Withdrawal by Subject | 56 | 49
Not completed — Lost to Follow-up | 1 | 4
Not completed — Received medication | 3 | 2
Not completed — Incomplete data | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Omega 3 and an Hypocaloric Diet: Participants will receive a supplement containing omega 3: DHA and EPA fatty acids together with an hypocaloric diet.
  Omega3 and an hypocaloric diet.: Thirty caps with the supplement will be provided every mo during three mo. Supplement will be administered as gel caps containing 1.1 g of DHA and EPA (®MaxEpa, Merck Laboratory) Hypocaloric diet will start at admission and will continue during the six months of follow-up. It will consist in providing a personalized diet including: a) reduction of 700 Kcal from the usual diet considering lipids and carbohydrates, b) increasing fruits and vegetables intake up to six portions daily each, and c) incrementing the intake of fiber to 30 g a day through the inclusion of whole grains.
- Total: Total of all reporting groups
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo | Total
Number analyzed (Participants) | 119 | 126 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 119 | 126 | 245
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.73 (1.97) | 13.58 (1.79) | 13.66 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 69 | 129
  Male | 59 | 57 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 119 | 126 | 245

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance
Description: Change from baseline in insulin resistance at three and six months. Changes in insulin resistance evaluated through Homeostasis Model Assessment Index (HOMA), calculated by formula: (glucose, mg * insulin,µU)/405. Where HOMA>3.16 indicated insulin resistance index.
Time Frame: At baseline (at diagnosis), three months, throughout six months.
Population: Of the participants analyzed at baseline and at month 3 (119 in omega 3 and an hypocaloric diet group and 126 Placebo group) only 80 and 82 participants respectively finished the study at month 6. The participants who did not finish the study, were because they did not want to take another blood sample at month 6.
Measure: Mean (Standard Deviation); unit: HOMA-IR Index
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
Number analyzed (Participants) | 119 | 126
HOMA-IR Index
  Homeostasis Model Assessment (HOMA) at baseline | 7.38 (4.21) | 6.89 (3.55)
  Homeostasis Model Assessment (HOMA) at 3 mo | 6.73 (3.71) | 6.28 (3.53)
  Homeostasis Model Assessment (HOMA) at 6 mo: number analyzed (Participants) | 80 | 82
  Homeostasis Model Assessment (HOMA) at 6 mo | 6.02 (3.21) | 5.41 (3.21)

2. Secondary Outcome: Nutritional Status
Description: Nutritional status was determined by registering body mass index (BMI) calculated by formula: kg/m^2.
Time Frame: At baseline (at diagnosis), three months, throughout six months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
Number analyzed (Participants) | 119 | 126
kg/m^2
  Body Mass Index at baseline | 31.53 (4.92) | 31.16 (3.79)
  Body Mass Index at 3 months | 30.89 (4.97) | 30.40 (3.79)
  Body Mass Index at 6 months: number analyzed (Participants) | 80 | 82
  Body Mass Index at 6 months | 31.1 (8.35) | 30.25 (3.95)

3. Other Pre Specified Outcome: Change in Insulin Resistance Through Fasting Insulin
Description: Change from baseline in insulin resistance at three and six months. Changes in insulin resistance evaluated through fasting insulin (µU/mL)
Time Frame: At baseline (at diagnosis), three months, throughout six months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
Number analyzed (Participants) | 119 | 126
µU/mL
  Fasting insulin at baseline | 33.05 (16.50) | 31.30 (15.05)
  Fasting insulin at 3 mo | 30.55 (15.52) | 29.09 (15.10)
  Fasting insulin at 6 mo: number analyzed (Participants) | 80 | 82
  Fasting insulin at 6 mo | 29.40 (12.57) | 27.23 (12.63)

4. Other Pre Specified Outcome: Nutritional Status Through Waist Circumference
Description: Nutritional status was determined by registering waist circumference in cm.
Time Frame: At baseline (at diagnosis), three months, throughout six months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
Number analyzed (Participants) | 119 | 126
cm
  Waist circumference at baseline | 100.44 (12.37) | 99.40 (9.81)
  Waist circumference at 3 months | 98.83 (12.33) | 97.66 (9.61)
  Waist circumference at 6 months: number analyzed (Participants) | 80 | 82
  Waist circumference at 6 months | 96.99 (11.68) | 97.11 (10.10)

ADVERSE EVENTS:
Arm/Group | Omega 3 and an Hypocaloric Diet | Placebo
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/126
Other Adverse Events (participants affected / at risk) | 0/119 | 0/126

LIMITATIONS AND CAVEATS:
We completed sample size at recruitment, but only 67% completed follow-up. We did not continue recruitment because preliminary analyses suggested that a huge sample size would be necessary to detect differences in insulin resistance (IR) and BMI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No